CLINICAL TRIAL: NCT05597631
Title: Does Adding Medium to Fresh Semen Samples Increase Motility After Preparation?
Brief Title: G-IVF and Sperm Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-GR-GIVFSP
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Infertility, Male
Keywords: Sperm motility; Sperm preparation; Osmolarity
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control
- G-IVF PLUS (Experimental): G-IVF PLUS
  Interventions: Device: G-IVF PLUS

INTERVENTIONS:
Device: G-IVF PLUS — Experimental
  Arms: G-IVF PLUS

SUMMARY:
The aim of this study is to investigate if adding a fixed volume of a physiological solution to a freshly produced sperm sample will affect sperm characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients producing a pre-clinical semen sample at the clinic

Exclusion Criteria:

* Patients with known azoospermia
* Patients who have had a vasectomy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 118 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of progressive motile sperm (%) | 10 minutes of assessment will be used to count the motile sperm for each sample.
  Proportion of progressive motile sperm after sample preparation

SECONDARY OUTCOMES:
Sperm yield (%) | 10 minutes used to assess motilty (as for primary outcome)
  Percentage of total number of motile sperm after sperm preperation

CONTACTS AND LOCATIONS:
Locations (1):
- IASO Maternity and Gynecology Clinic, Marousi, Greece